CLINICAL TRIAL: NCT01858142
Title: Preparing Parents to be Present for Their Child's Anesthesia Induction: A Randomized Control Effectiveness Trial
Brief Title: Helping Parents to Decide Whether They Want to be With Their Child During Anesthesia Induction
Acronym: PPDT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IWK Health Centre (Other)
Responsible Party: Principal Investigator, Patrick J. McGrath, Supervisor, IWK Health Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1012940
Record Dates: First submitted 2013-05-09; First posted 2013-05-21 (Estimated); Last update posted 2016-03-21 (Estimated); Status verified 2016-03

CONDITIONS: Pre-operative Anxiety
Keywords: Pediatric anesthesia; Pre-operative anxiety; parental presence; children; elective surgical procedures; mask induction
MeSH Terms: interventions — Reference Standards

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Preparation intervention (Experimental): The parental presence decision tool will be delivered as an App shown to families using an iPAD and a set of headphones. This App will include information on what to expect in the operating room as well as the role of the parents. The App incorporates the basic principles of other effective perioperative preparation interventions (e.g., providing both sensory and procedural information) and is tailored to the local context. In addition to preparatory information, the App will also inform parents of the role of parent anxiety on children's outcomes in the operating room.
  Interventions: Behavioral: Parental presence decision tool
- Standard preparation (Placebo Comparator): In standard preparation condition, treating nurses and anesthesiologists will provide information to parents as they standardly do when parents are present at induction; this includes information on logistical issues and safety in the operating room (e.g., where to stand, how to put on gown) and risks of anesthesia induction. Additionally, parents in the standard preparation condition will view a summary of this standard information as text on an iPAD.
  Interventions: Behavioral: Standard preparation

INTERVENTIONS:
Behavioral: Parental presence decision tool
  Arms: Preparation intervention
Behavioral: Standard preparation
  Arms: Standard preparation

SUMMARY:
Children are distressed at anesthesia induction and this distress can result in maladaptive recovery outcomes. Having parents be present at anesthesia induction (PPIA) has been suggested as a potential intervention to decrease children's distress, and this intervention is widely favored by parents. However, to date, PPIA has not been found to be effective in reducing children's anxiety. The lack of efficacy may be attributable to the fact that parents have generally not been prepared for PPIA. The one study that prepared parents (as part of a larger preoperative preparation program) found that PPIA with preparation was superior to PPIA as previously studied (without preparation). Unfortunately, this program is resource intensive and therefore is not clinically feasible. This study will compare PPIA with a clinically feasible preparation program to PPIA with standard care (minimal preparation). Should our intervention show evidence of efficacy, the investigators will have designed a program that is easily translatable to everyday clinical practice. This will, in turn, reduce children's anxiety, improve postoperative outcomes and increase parental satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Ages 2 to 10
* Scheduled for elective surgical procedure at IWK Health Centre
* Mask induction
* ASA classification I or II

Exclusion Criteria:

* Intravenous induction
* Diagnosed development delay
* ASA classification III or higher
* Pre-medication with benzodiazepine

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 104 (Actual)
Dates: Start 2013-06; Primary Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Modified Yale Pre-Operative Anxiety Scale | post-treatment (following intervention); average=15 minutes after treatment
  Yale Preoperative Anxiety Scale (mYPAS; Kain et al., 1997). This researcher completed measure is made up of 5 categories (e.g., activity, vocalizations) each rated on ordinal behaviorally anchored scales. Total scores on the measure range from 23 to 100, with higher scores indicating higher child anxiety at induction. The tool has shown good convergent validity with another measure of child anxiety (r = 0.79), and excellent inter-rater reliability (kappa range 0.63-0.90). A cutoff score of 30 has been shown to have the best balance of sensitivity (0.85) and specificity (0.92).
  NOTE: Most of the measure is administered post-treatment, but part of it begins pre-treatment at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Jill Chorney, PhD, Principal Investigator — IWK Health Centre
Locations (1):
- IWK Health Centre, Halifax, Nova Scotia, Canada